CLINICAL TRIAL: NCT07285200
Title: Examining the Care Burden of Caregivers of Peritoneal Dialysis Patients Using the Q Method
Brief Title: Care Burden in Peritoneal Dialysis Caregivers.
Status: Completed | Type: Observational
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Yavuz Uren, Principal Inverstigator, Yuzuncu Yil University
Other Study IDs: PD-Q1
Record Dates: First submitted 2025-11-18; First posted 2025-12-16 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Peritoneal Dialysis
Keywords: Caregivers; Q methodology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aimed to explore the subjective opinions and perspectives of peritoneal dialysis caregivers regarding the caregiver burden they experience.

DETAILED DESCRIPTION:
Caregiving significantly contributes to the development of caregiver burden in caregivers of peritoneal dialysis patients. This study aimed to explore the subjective opinions and perspectives of peritoneal dialysis caregivers regarding the caregiver burden they experience. This study was conducted using the Q methodology because it allows working with small sample sizes.

ELIGIBILITY:
Inclusion Criteria:

* Must be between 18 and 65 years of age,
* Must be able to read and write,
* Must have no vision or hearing problems,
* Must be willing to participate in our study,
* Must be conscious and have no psychiatric problems,
* Must have no communication problems,
* Must be related to the patient.

Exclusion Criteria:

* Lack of a permanent caregiver (constant change),
* Desire to leave the job.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: There are 12 peritoneal dialysis patients in the province where the study was conducted. The goal was to reach the entire population, but only nine caregivers were reached. Q methodology was preferred because it allows for small sample sizes.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2025-04-20 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Subjective views of caregivers survey | up to 6 months
  Subjective views of caregivers of peritoneal dialysis patients regarding care burden

CONTACTS AND LOCATIONS:
Overall Officials: YAVUZ UREN, Dr., Study Director — yavuzuren@yyu.edu.tr
Locations (1):
- Sbu. Van Training and Research Hospital, Van, Turkey (Türkiye)